CLINICAL TRIAL: NCT06120023
Title: Post-Market Clinical Follow Up for Total Knee Arthroplasty System Madison
Acronym: 2022-07
Status: Recruiting | Type: Observational
Sponsor: Societe dEtude, de Recherche et de Fabrication (Industry)
Responsible Party: Sponsor
Other Study IDs: 2022-07_Madison3
Record Dates: First submitted 2023-10-18; First posted 2023-11-07 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Knee Arthropathy
Keywords: total knee prosthesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
MADISON Total Knee Prosthesis is intended to be used for total knee arthroplasty to reduce pain and restore joint mobility of the knee.

Clinical data for MADISON Total Knee Prosthesis available are not deemed sufficient to support performance and benefits claimed on the whole lifetime of the product.

Thus, in order to maintain compliance with the EU regulation (2017/745) related to medical devices and following ISO 14/155:2020, SERF has set up post-market clinical follow-up study (PMCF) to confirm safety and performance of Total Knee Arthroplasty system MADISON. This study is designed to cover the expected 15-years follow-up, to retrieve data according to implant feature (Posterior Stabilized or Ultra Congruent) or fixation method and to gather data related to the revision of partial knee prosthesis.

The primary objective of this study is to assess the clinical safety of MADISON total knee prostheses. The secondary objective is to evaluate the survival rates, the clinical performances and clinical benefits of MADISON total knee prosthesis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults (≥ 18 years) covered by French social security system
* Diagnosed with:

  * Osteoarthritis (primary and secondary),
  * Revision of a unicompartmental knee prosthesis.
* Patient requiring a surgery and implantation of a Madison TKA (Total Knee Arthroplasty)
* Patient physically and mentally able to comply with protocol, meet the follow-up visits as deemed by the investigator and fill in quality of life questionnaire.
* Patient having signed a written informed consent

Exclusion Criteria:

* Progressive, acute or chronic infection, local to the operative site or systemic that may affect the prosthetic joint,
* Any loss of musculature or serious lesions of muscles, nerves and/or blood vessels deficiency, putting the affected limb at risk,
* Lack of bone substance or inadequate bone quality on femoral or tibial surfaces, as it might compromise the stability of the prosthesis components,
* Skeletal immaturity,
* Pathologies that may compromise the functionality of the implant in any way (i.e. osteomyelitis, neuropathic joint),
* Parameters incompatible with satisfactory long-term results (i.e. age, weight,
* Neurological condition of the patient incompatible with the post-operative constraints associated with this type of intervention,
* Known allergy to one of the implant components.
* Severe obesity with or without comorbidities
* Pregnant or nursing women,
* Patients with a contraindication to radiography
* Patients deprived of their liberty or hospitalised without their consent
* Patients under legal protection (e.g. guardianship)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subjects with a diagnosis of knee replacement surgery requiring to be implanted with a TKA (Total Knee Arthroplasty) system MADISON according to instructions for use. Patients will be followed according to current practice.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-10-17 (Actual); Primary Completion 2040-12-31 (Estimated); Study Completion 2040-12-31 (Estimated)

PRIMARY OUTCOMES:
Revision rate according to Kaplan-Meier | 15 years
  Assess the revision rate, whatever the cause of revision, including infection at 15 years

SECONDARY OUTCOMES:
Survival rate according to Kaplan-Meier | From per operative period to 15 years
  Assess the survival rate, whatever the cause of revision, including infection at 1 year, 3 years, 5 years and 10 years follow-up
Adverse events | From per operative period to 15 years
  List type and occurence of adverse events
Functional improvement using 2011KSS score | From per operative period to 15 years
  2011 KSS stands for Knee Society Score Assessement of functional improvement picked up from global 2011KSS score. The functional score is composed of four subgroups and is rating from 0 to 100 (higher score means a better outcome).
Patient's expectation / satisfaction using 2011KSS score | From per operative period to 15 years
  2011 KSS stands for Knee Society Score Evaluation of patient's expectation / satisfaction is picked up from global 2011KSS score.
  This evaluation is rating from 0 to 55 (higher score means a better outcome).
Pain reduction using 2011KSS score | From per operative period to 15 years
  2011 KSS stands for Knee Society Score Pain reduction evaluation is picked up from the symptom score of global 2011KSS score.
  This score is rating from 0 to 25 (higher score means a better outcome).
Pain Evaluation using KOOS | From per operative period to 15 years
  Evaluate pain using KOOS score. KOOS stands for Knee Injury and Osteoarthritis Outcome Score. The questionnaire has five separately scored subscales: Pain, Function in Daily Living (ADL), Function in Sport and Recreation, Other Symptoms, and Knee-Related Quality of Life (QOL).
  Pain evaluation is picked up from global KOOS score. Each question is assigned a score (0-4) and a normalized score is calculated for each subscale (100 indicates no symptoms and 0 indicates extreme symptoms)
Functional improvement in Daily Living using KOOS | From per operative period to 15 years
  Evaluate Function in Daily Living (ADL) using KOOS score. KOOS stands for Knee Injury and Osteoarthritis Outcome Score. The questionnaire has five separately scored subscales: Pain, Function in Daily Living (ADL), Function in Sport and Recreation, Other Symptoms, and Knee-Related Quality of Life (QOL).
  Function in Daily Living (ADL) evaluation is picked up from global KOOS score. Each question is assigned a score (0-4) and a normalized score is calculated for each subscale (100 indicates no symptoms and 0 indicates extreme symptoms)
Functional improvement in Sport and Recreation using KOOS | From per operative period to 15 years
  Evaluate Function in Sport and Recreation using KOOS score. KOOS stands for Knee Injury and Osteoarthritis Outcome Score. The questionnaire has five separately scored subscales: Pain, Function in Daily Living (ADL), Function in Sport and Recreation, Other Symptoms, and Knee-Related Quality of Life (QOL).
  Function in Sport and Recreation evaluation is picked up from global KOOS score.
  Each question is assigned a score (0-4) and a normalized score is calculated for each subscale (100 indicates no symptoms and 0 indicates extreme symptoms)
Functional improvement Other Symptoms using KOOS | From per operative period to 15 years
  Evaluate Other Symptoms using KOOS score. KOOS stands for Knee Injury and Osteoarthritis Outcome Score. The questionnaire has five separately scored subscales: Pain, Function in Daily Living (ADL), Function in Sport and Recreation, Other Symptoms, and Knee-Related Quality of Life (QOL).
  Other Symptoms evaluation is picked up from global KOOS score. Each question is assigned a score (0-4) and a normalized score is calculated for each subscale (100 indicates no symptoms and 0 indicates extreme symptoms)
Assessement of Knee-Related Quality of Life using KOOS | From per operative period to 15 years
  Evaluate Knee-Related Quality of Life (QOL) using KOOS score. KOOS stands for Knee Injury and Osteoarthritis Outcome Score. The questionnaire has five separately scored subscales: Pain, Function in Daily Living (ADL), Function in Sport and Recreation, Other Symptoms, and Knee-Related Quality of Life (QOL).
  Knee-Related Quality of Life (QOL) assessement is picked up from global KOOS score.
  Each question is assigned a score (0-4) and a normalized score is calculated for each subscale (100 indicates no symptoms and 0 indicates extreme symptoms)
Oblivion of prosthesis | From per operative period to 15 years
  Assess the degree of forgetfulness of the prosthesis using FJS-score (Forgotten Joint Score):
  FJS stands for Forgotten Joint Score. The Forgotten Joint Score assessement consists of 12 questions and is scored on a 0-100 scale. The higher is the score, the less the patient is aware of their affected joint when performing daily activities.
Mobility improvement | From per operative period to 15 years
  Assessed by the surgeon through questionary with a 4 item-scale : significant improvement / slight improvement / identical mobility / decrease of mobility

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique de la Sauvegarde, Lyon, Rhône, France